CLINICAL TRIAL: NCT05233553
Title: High Incidence of Secondary Sclerosing Cholangitis in Hospitalized "First-wave" COVID-19 Patients: a Retrospective Single Center Study
Brief Title: SSC-COVID in Patients After COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 431/2020BO
Record Dates: First submitted 2022-02-09; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2020-02

CONDITIONS: Secondary Sclerosing Cholangitis; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- post-COVID-patients
  Interventions: Other: control of liver enzymes

INTERVENTIONS:
Other: control of liver enzymes — follow-up with clinical and laboratory measurements

SUMMARY:
Analysis of occurrence of SSC-COVID in SARS-CoV-2-patients after the first wave of COVID-pandemic

DETAILED DESCRIPTION:
In Central Europe, the first wave of SARS-CoV-2 peaked in April 2020 and ended in June 2020. Our tertiary care center, the University Hospital of Tübingen is located in a first-wave SARS-CoV-2 hotspot area that had the second highest 7-day incidence in Germany on March 31, 2020, exactly at the peak of the first wave in Germany (205.9/100,000, www.rki.de; the peak daily incidence in Tübingen was 179/100,000 on March 25, 2020). In this period, 249 patients were hospitalized for or with SARS-CoV-2 infection.

To gain fast knowledge about the new disease, a COVID-19 patient registry was established at our center, including all patients admitted to Tübingen University Hospital for or with SARS-CoV-2 infection and retrospectively collecting routine clinical data. After hospitalization, patients were followed up in the outpatient clinic of our department, the Department of Gastroenterology, Hepatology, Gastrointestinal Oncology, Geriatrics and Infectious Diseases.

Subsequently, several patients with secondary sclerosing cholangitis (SSC) after COVID-19 (SSC-COVID) were recognized in our center, either from our own cohort, or referred to our center due to the need for further treatment of end-stage liver disease including liver transplantation. SSC is a cholangiopathy estimated to be rare in ICU patients with an incidence of 1/2000 ICU patients. Pathogenesis has not been fully deciphered, but a combination of ischemic injury and increased bile toxicity during critical illness is suspected. This imposes acute damage on the biliary system, that, if not resolving early or spontaneously, may lead to the vicious circle of gradually destruction of the biliary tree over time, well known to hepatologists and endoscopists.

ELIGIBILITY:
Inclusion Criteria:

* post-COVID19-patients with required hospitalization during the first wave of COVID-19-pandemic
* patients controlled at the university ambulance for follow-up

Exclusion Criteria:

* children and patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a study of adult patients who participated in the COVID-19 outpatient clinic at the University Hospital of Tübingen as part of the follow-up examinations after COVID-19 disease. In particular, the development of liver enzymes was analysed.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of SSC-COVID in hospitalized COVID-patients of the first wave | one and a half year
  While Follow-up-session controlled clinical and laboratory parameters

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided
IPD are anonymised, the consent has been obtained from the ZKS.